CLINICAL TRIAL: NCT03558256
Title: The Study of Mindfulness-based Cognitive Therapy and Major Depressive Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MBCT2018
Record Dates: First submitted 2018-05-30; First posted 2018-06-15 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-05

CONDITIONS: Major Depressive Disorder
Keywords: Mindfulness-Based Cognitive Therapy
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Mindfulness-Based Cognitive Therapy; Dosage Forms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based Cognitive Therapy (Experimental): MBCT group is a treatment group used mindfulness- based cognitive therapy added to the usual medication treatment, and guided by two therapists for 8 sessions. Every group of 6 people can form a closed structural group. Each session lasts 2 hours once a week, and has daily homework assignments.
  Interventions: Behavioral: Mindfulness-based Cognitive Therapy; Drug: Medication
- Medication (Active Comparator): Medication group is a control group that can choose to use the serotonin reuptake inhibitors (SSRIs) approved by China food and Drug Administration (SFDA) for the treatment of depression (fluoxetine, paroxetine, fluvoxamine, sertraline, citalopram and escitalopram).
  Interventions: Drug: Medication

INTERVENTIONS:
Behavioral: Mindfulness-based Cognitive Therapy — Patients participating in the experimental group will receive the MBCT intervention besides the usual medication treatment. The intervention is implemented by the manual adapted from the MBCT for Depression (Segal et al. 2013). The modified version of the program has the same structure with the original manual combined the mindfulness training and the cognitive elements from CBT, but the content is more suitable for the Chinese. The instructors in this study are trained and certificated psychiatrists and psychotherapists with rich experience of working with MDD, and they will receive a weekly supervision conducted by a senior supervisor.
  Arms: Mindfulness-based Cognitive Therapy
Drug: Medication — Both of the MBCT group and the medication group will receive the medication treatment. The initial dose conforms the drug instructions, the dosage can be adjusted once a week, and the maximum dosage should not exceed the maximum amount by the instructions. MDD patients with sleep disorders can use drugs combined with benzodiazepine drugs, but not continuing for more than two weeks; while other psychotropic drugs are not allowed. All of the drugs used in this study are usual clinical drugs with good security, the common adverse reactions include nausea, dry mouth, constipation, diarrhea, indigestion, dizziness, drowsiness, fatigue, sweating, heart palpitations, delayed ejaculation in male, increasing blood aminotransferase without symptoms occasionally and so on.

SUMMARY:
The primary objective of the study is to evaluate the clinical curative effect of mindfulness-based cognitive therapy(MBCT) for major depressive disorder(MDD). Moreover, we will also explore the relationship between P300 potential and erroneous negative potential (ERN) variation and clinical symptoms in MDD and MBCT.

This study is a randomized-control trial with two study arms: half of patient cases will receive usual medication treatment with the serotonin reuptake inhibitors (SSRIs) and half of patient cases will receive MBCT added to the usual medication treatment. This study is also a case-control trial, there will be matched normal controls compared with patient cases through a range of psychological scales and electroencephalogram.

DETAILED DESCRIPTION:
The study is designed as a prospective, assessor-blinded, randomized-control, case-control clinical trial with 70 MDD cases and 35 matched normal controls.After signed the Informed consents, MDD cases will be assigned to two groups randomly by the table generated by Microsoft Excel 2010 to ensure the random distribution between groups. The group of each patient will be allotted by the research coordinator so that evaluators will be blind about it, and patients will be asked to not mention the intervention conditions to evaluators.

As the research tools, a range of self-rating scales, other-rating scales and behavioral tests and EEG will be mainly applied to assess clinical symptoms and brain state of participants at baseline (week 0), during the intervention (week 2, 4 and 6), at the end of the intervention (week 8), and during the maintenance phase (week 12, 20 and 32).

After 8-week intervention, all of the participants including MDD cases and normal controls will enter the follow-up. Participants of medication group will continue their treatment options without changing the types and doses of medication compared with what they used in the intervention period. MBCT group is the same that participants will maintain their medication treatment and practice MBCT exercises at home.

ELIGIBILITY:
Inclusion criteria for patient cases:

* Male or female, age between 18-55 years.
* Junior/middle school education or above.
* Meet the DSM- IV diagnosis of MDD by the evaluation of Chinese version of M.I.N.I. and the clinical diagnosis of one associate chief and above psychiatrist.
* HAMD24 score ≥ 8.
* Have not yet accepted psychiatric medication, or had received irregular medication treatment and had discontinued it for 8 weeks.
* Have enough visual and acoustic ability to complete the inspection required for the study.
* Each patient should be willing to participate in this study, he/she and his/her guardian must sign the informed consent form after understanding the nature of this study.

Inclusion criteria for normal controls:

* Healthy population matched patient cases in age, sex and education; Male or female; age between 18-55 years; Junior/middle school education or above.
* Excluded the possibility of mental disorders by the evaluation of Chinese version of M.I.N.I. and the psychiatric interview of one associate chief and above psychiatrist.
* HAMD24 score < 8; HAMA score < 7.
* No psychotropic drug history.
* No history of two lines of three generations of mental disorders.
* Have enough visual and acoustic ability to complete the inspection required for the study.
* Each patient should be willing to participate in this study, he/she and his/her guardian must sign the informed consent form after understanding the nature of this study.

Exclusion criteria for patient cases:

* Meet DSM-IV Axis I disorder diagnostic criteria for other psychiatric disorders.
* Have severe depression symptoms (HAMD24 score > 35), psychotic symptoms, negative self-concept or a risk of suicide.
* Persons with severe physical disease or central nervous system disease, and with substance abuse.
* Pregnancy or ready to be pregnant and lactating women.
* Had previously received systematic MBCT intervention, with no significant effect.

Exclusion criteria for normal controls:

* Have negative self-concept or a risk of suicide.
* Persons with severe physical disease or central nervous system disease, and with substance abuse.
* Pregnancy or ready to be pregnant and lactating women.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Estimated)
Dates: Start 2016-05-16 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of Hamilton Depression Scale-24 from baseline to 32 weeks | baseline (week 0), during the treatment (week 2, 4, 6), end of treatment (week 8), and during the maintenance phase (weeks 12, 20 and 32)
  The Hamilton Depression Scale-24 (HAMD-24) is the most common other-rating scale to measure the severity of depression symptoms for adult. It is a clinical instrument with good validity and reliability, and most of the 24 items weighted from 0 to 4.

SECONDARY OUTCOMES:
Change of Hamilton Anxiety Scale from baseline to 32 weeks | baseline (week 0), during the treatment (week 2, 4, 6), end of treatment (week 8), and during the maintenance phase (weeks 12, 20 and 32)
  The Hamilton Anxiety Scale (HAMA) is a common clinician-administered scale to measure the state of anxiety among adults with anxiety symptoms. There are 14 items of the 5-point rated scale.
Change of Self Compassion Scale from baseline to 32 weeks | baseline (week 0), during the treatment (week 2, 4, 6), end of treatment (week 8), and during the maintenance phase (weeks 12, 20 and 32)
  The Self Compassion Scale (SCS) is proved to be an instrument featured good characteristics for reliability and validity. There are 26 items divided into 6 Subscales (out of 5 points from almost never to almost always), including self-kindness, self-judgment, common humanity, isolation, mindfulness and over-identification.

CONTACTS AND LOCATIONS:
Overall Officials: Yifeng Shen, Senior, Study Director — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zhang T, Wang L, Bai Y, Zhao W, Wu Y, Jiang W, Fan Q, Qiu J. Mindfulness-Based Cognitive Therapy in Major Depressive Disorder: A Study Protocol of a Randomized Control Trial and a Case-Control Study With Electroencephalogram. Front Psychiatry. 2021 Jul 26;12:499633. doi: 10.3389/fpsyt.2021.499633. eCollection 2021. PMID 34381382